CLINICAL TRIAL: NCT01875523
Title: A Single Dose, Open-label, Parallel-group Study to Assess the Pharmacokinetics of Serelaxin in Patients With Severe Renal Impairment or End-Stage Renal Disease on Hemodialysis Compared to Matched Healthy Control Subjects
Brief Title: PK of Serelaxin in Severe Renal Impairment and ESRD
Acronym: CRLX030A2102
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CRLX030A2102; 2013-001875-18 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-12 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2014-04

CONDITIONS: Renal Failure, Chronic; End-Stage Renal Disease
Keywords: Renal disease; renal impairment; End stage renal disease; Healthy volunteer; Pharmacokinetics
MeSH Terms: conditions — Kidney Failure, Chronic; Kidney Diseases; Renal Insufficiency | interventions — serelaxin protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 Treatment with serelaxin (Experimental): Patients with severe renal impairment will receive a single 4 hour i.v. infusion of serelaxin
  Interventions: Drug: Serelaxin
- Group 2 Treatment with serelaxin (Experimental): Patients with end stage renal disease will receive a single 4 hour i.v. infusion of serelaxin and dialysis will be done on the day of treatment
  Interventions: Drug: Serelaxin
- Group 3 Treatment with serelaxin (Experimental): Patients with end stage renal disease will receive a single 4 hour i.v. infusion of serelaxin and treatment and PK will be done in dialysis-free interval
  Interventions: Drug: Serelaxin
- Group 4 Treatment with serelaxin (Experimental): Healthy volunteers will receive a single 4 hour i.v. infusion of serelaxin and dialysis will be done on the day of treatment
  Interventions: Drug: Serelaxin

INTERVENTIONS:
Drug: Serelaxin
  Other Names: RLX030

SUMMARY:
The study is designed to evaluate the pharmacokinetics, safety and tolerability, immunogenicity and pharmacogenetics of a single dose of serelaxin/RLX030 in patients with severe renal impairment and end-stage-renal-disease (ESRD) compared to healthy volunteers.

ELIGIBILITY:
Inclusion criteria:

All subjects

- at least 50 years; body mass index (BMI) within the range of 18 - 35 kg/m2.

Patients with severe renal impairment / ESRD

* Severe renal impairment (clinically significantly abnormal creatinine and creatinine clearance (15mL/min/1.73m2≤eGFR<30mL/min/1.73m2) or ESRD on hemodialysis.
* Sitting vital signs should be within the following ranges:
* oral body temperature between 35.0-37.5 °C
* systolic blood pressure, 110 to 170 mm Hg
* diastolic blood pressure, 60 to 105 mm Hg
* pulse rate, 45 - 100 bpm

Healthy subjects

* eGFR > 90mL/min/1.73m2;
* matching in race, age (±10 years), gender, BMI (±15%) to a subject with renal impairment
* Subject must be in good health.
* Sitting vital signs should be within the following ranges:
* oral body temperature between 35.0-37.5 °C
* systolic blood pressure, 100 to 150 mm Hg
* diastolic blood pressure, 60 to 95 mm Hg
* pulse rate, 50 to 100 bpm

Exclusion Criteria:

All subjects

* History of clinically significant ECG abnormalities at Screening or Baseline.
* Pregnant or nursing (lactating) women
* Women of child-bearing potential unless they are using highly effective methods of contraception during dosing of study treatment.
* Sexually active males (incl. vasectomized men) must use a condom during intercourse while taking drug and for 2 weeks after stopping study medication.
* Recent (within the last three years) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).

Patients with severe renal impairment / ESRD:

* Presence of any non-controlled and clinically significant disease, surgical or medical condition that could affect the study outcome or that would place the patient at undue risk as judged by the investigator.
* Hemoglobin levels below 9.0 g/dL at screening and baseline, other laboratory parameters at screening and baseline outside acceptable limits .
* Treatment with any cytostatic drug or autonomic alpha blocker.

Healthy subjects:

* Use of any prescription drugs (other than hormonal contraception, herbal supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing.
* History or presence of any disease, surgical or medical condition of any major system organ class considered clinically significant by the investigator.
* Laboratory parameter at screening and baseline outside of normal limits. For small deviations which could be attributed to the characteristics of the subjects (e.g. age) it will be to the discretion of the investigator to consider them as exclusive or not.
* A positive Hepatitis B surface antigen or Hepatitis C test result.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (AUClast) | pre-treatment, 15 min, 1, 2, 3, 4, 4:15, 5, 6, 7, 8, 9, 10, 12, 24, 28, 36, 48 hours and day 15
  Blood samples will be collected on days 1 through 3 and then on Day 15 for the determination of serum concentrations of serelaxin
The area under the serum concentration-time curve from time zero to 28 hours after administration (AUC 0-28hr) | pre-treatment, 15 min, 1, 2, 3, 4, 4:15, 5, 6, 7, 8, 9, 10, 12, 24, 28, 36, 48 hours and day 15
  Blood samples will be collected on days 1 through 3 and then on Day 15 for the determination of serum concentrations of serelaxin
The area under the serum concentration-time curve from time zero to infinity (AUCinf) | pre-treatment, 15 min, 1, 2, 3, 4, 4:15, 5, 6, 7, 8, 9, 10, 12, 24, 28, 36, 48 hours and day 15
  Blood samples will be collected on days 1 through 3 and then on Day 15 for the determination of serum concentrations of serelaxin
The observed maximum serum concentration following drug administration (Cmax) | pre-treatment, 15 min, 1, 2, 3, 4, 4:15, 5, 6, 7, 8, 9, 10, 12, 24, 28, 36, 48 hours and day 15
  Blood samples will be collected on days 1 through 3 and then on Day 15 for the determination of serum concentrations of serelaxin

SECONDARY OUTCOMES:
Percentage of patients with reported adverse events, serious adverse events and death. | From Day -21 to Day 15
Percentage of patients developing anti-RLX030 antibodies | Day 1 (pre-treatment) and Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Grünstadt, Germany

REFERENCES:
- See also: Results for CRLX030A2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13044